CLINICAL TRIAL: NCT00105781
Title: Nurse Physical Activity Counseling in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRI 99-334
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-05

CONDITIONS: Frail Elderly; Aged; Physical Fitness
Keywords: Nurses; Telephone; Counseling; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Exercise counseling

INTERVENTIONS:
Behavioral: Exercise counseling

SUMMARY:
Aging veterans with functional impairments followed in primary care clinics were randomized to counseling for a walking plus strength exercise home-based exercise program or to health education by a nurse. Exercise participants attended 3 intervention sessions totaling about 100 minutes of contact with the nurse and a physical therapy assistant over 10 months. They were also asked to record walking and strength exercise on monthly calendars and received motivational automated phone messages. Education control patients discussed health topics of their choice with the nurse. Materials were based on National Institute of Aging materials currently available on the internet. After 10 months, the exercise participants reported more time spent in walking and strength exercise and accelerometer data indicated a greater increase in time spent in moderate or higher intensity activity per day. Participants who engaged in strength exercises improved more on functional fitness tests and quality of life after 10 months. Analyses from the cognitive sub-study remain incomplete.

DETAILED DESCRIPTION:
Description Background: Many older individuals are at high risk for health complications and functional impairment due to low levels of physical activity. Walking is an acceptable and safe activity associated with many health benefits. Strength and flexibility exercises are also important components of the exercise prescription for optimal health and function in the elderly. Developing interventions to promote healthy physical activity is a current public health priority, and counseling by providers in health care settings is a promising approach. Objectives: The primary objective was to evaluate the effects of nurse counseling on total weekly minutes and frequency of home-based walking and strength/flexibility exercises. Secondary objectives included evaluating physical function and accelerometer physical activity. A sub-study initiated in April 2004 examined the association between exercise and cognitive functioning. Methods: The design is a randomized clinical trial. Outcomes were assessed at 5 months (end of initiation phase) and 10 months (maintenance). Clinic-based exercise counseling was delivered by a nurse and physical therapy assistant at baseline and a 1-month follow-up. Interventions were based on exercise for people over 50 information available on the National Institute on Aging internet website. VA primary care patients aged 60 to 85 referred by their primary care provider were assigned to one of 2 conditions: a) exercise counseling or b) health education contact control. All participants received preventive health counseling emphasizing safety and falls prevention. The exercise counseling group also received follow-up phone contacts, including automated motivational messages, from the nurse. All participants had continuing contact with research staff but were exposed to different specific intervention components. . Status: Data collection complete; additional analyses in progress.

ELIGIBILITY:
Inclusion Criteria:

Referred by primary care providers in VA primary care clinics. Interested and willing to try to increase physical activity. Some self-reported or observed impairments in physical function. Excluded if there are health conditions that make home-based exercise not appropriate. Observed or self-reported physical function impairment Able to walk for health Living independently in community Able to return to VA MedicalCenter for research visits Enrolled in primary care Access to telephone

Exclusion Criteria:

Any of these within 6 months: myocardial infarction, congestive heart failure, TIA or stroke, leg fracture, seizure, uncontrolled arrhythmia, unstable angina Uncontrolled diabetes, hypertension, dyslipidemia FEV1 less than 1.5 Any condition that provider believes would make unsupervised exercise unsafe

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2002-11; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Minutes and days per week of walking and strength training exercise at 5 and 10

SECONDARY OUTCOMES:
Functional fitness tests, Accelerometer activity, Quality of Life, and Cognitive performance in sub-sample

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. Dubbert, PhD, Principal Investigator — G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS
Locations (1):
- G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS, Jacksonport, Arkansas, United States

REFERENCES:
- [Result] Dubbert PM, Morey MC, Kirchner KA, Meydrech EF, Grothe K. Counseling for home-based walking and strength exercise in older primary care patients. Arch Intern Med. 2008 May 12;168(9):979-86. doi: 10.1001/archinte.168.9.979. PMID 18474762